CLINICAL TRIAL: NCT05966883
Title: SpermQT Prospective Observational Trial
Acronym: SPOT
Status: Recruiting | Type: Observational
Sponsor: Inherent Biosciences (Industry)
Collaborators: Yale University (Other); Boston IVF (Other); Shady Grove Fertility (Unknown); University of Washington (Other); Brigham Young University (Other); Male Fertility and Sexual Medicine Specialists (Unknown); Inception Fertility Research Institute, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SPOT001
Record Dates: First submitted 2023-05-30; First posted 2023-08-01 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Male Infertility
Keywords: Epigenetics
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to validate the ability of the Epigenetic Sperm Quality Test (SpermQT) to assess a man's sperm quality and corresponding success of infertility treatments.

DETAILED DESCRIPTION:
This prospective study will consist of analyzing a man's semen sample to determine the patient's SpermQT score and following the success of each fertility treatment to produce a pregnancy and live birth. Physicians and patients will be blinded to SpermQT results.

ELIGIBILITY:
Inclusion Criteria:

* The subjects have been recommended to pursue IUI, or they have recently completed an IUI (regardless of outcome)
* Male partner is under 45 years of age
* Female partner is under 38 years of age
* The total motile sperm count from the raw semen analysis must be greater than or equal to 10 million

Exclusion Criteria:

* The female or male partner have a BMI equal to or greater than 40
* The male partner has undergone male testosterone replacement therapy in the last 6 months
* Either the female or male partner have a history of recurrent pregnancy loss, defined as 2 or more consecutive clinical/ultrasound pregnancy losses
* There are any known factors contributing to female factor infertility, such as but not limited to:
* Severe Endometriosis (stage 3 or higher, endometrioma on ovaries)
* Multiple uterine fibroids 5cm or larger
* Severe Asherman's Syndrome
* Severe Mullerian anomaly
* Lack of tubal patency in at least one fallopian tubes

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Couples that are eligible for an IUI procedure and/or have been recommended to pursue IUI, and/or couples have recently completed an IUI cycle (no matter the outcome)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that have and have not achieved pregnancy during rounds 1 and 2 of intrauterine insemination (IUI) | 6 months
  Number of patients that have and have not achieved pregnancy during rounds 1 and 2 of IUI in each bracket of SpermQT score (Poor, Normal, and Excellent)

SECONDARY OUTCOMES:
Number of patients that have and have not achieved pregnancy during subsequent rounds of intrauterine insemination (IUI) and in vitro fertilization (IVF) | 18 months
  Number of patients that have and have not achieved pregnancy during subsequent rounds of IUI and with IVF in each bracket of SpermQT score (Poor, Normal, and Excellent)
Number of patients that have and have not achieved a live birth | 18 months
  Number of patients that have and have not achieved a live birth in each bracket of SpermQT score (Poor, Normal, and Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Brogaard, PhD, Principal Investigator — Inherent Biosciences
Locations (6):
- United States (6):
  - Male Fertility and Sexual Medicine Specialists, San Diego, California
  - Shady Grove Fertility, Greenwood Village, Colorado
  - Yale Medicine, Orange, Connecticut
  - Boston IVF, Waltham, Massachusetts
  - Inception Fertility, LLC, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No